CLINICAL TRIAL: NCT06040957
Title: Bone Marrow vs Adipose Tissue as a Cell Source for Infiltrative Treatment of Knee Osteoarthritis: Randomized Clinical Trial
Brief Title: Bone Marrow Versus Adipose Tissue as a Cell Source for Infiltrative Treatment of Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAST-GR
Record Dates: First submitted 2023-08-09; First posted 2023-09-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: bone marrow aspirate concentrate; minimally manipulated adipose tissue; BMAC; MM-AT; intra-articular injection; knee injection; mesenchymal stromal cells; Randomized controlled trial; cellular orthobiological products
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This is a randomized trial with 1:1 allocation.
Who Masked: Outcomes Assessor
Masking Description: To ensure the blinding of the health care personnel who will perform the checks (single-blind), follow-up visits will be performed by physicians not involved in the treatment procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single intra-articular injection of BMAC (Experimental): Patients randomized in this group will undergo single knee intra-articular injection of bone marrow aspirate concentrate (BMAC)
  Interventions: Biological: Bone marrow aspirate concentrate injection
- single intra-articular injection of MM-AT (Experimental): Patients randomized in this group will undergo single knee intra-articular injection of minimally manipulated adipose tissue (MM-AT)
  Interventions: Biological: intra-articular injection of Minimally manipulated adipose tissue

INTERVENTIONS:
Biological: Bone marrow aspirate concentrate injection — single intra-articular injection of Bone Marrow aspirate concentrate derived from the patient's iliac crest
  Arms: single intra-articular injection of BMAC
Biological: intra-articular injection of Minimally manipulated adipose tissue — single intra-articular injection of Minimally manipulated adipose tissue derived from the patient's abdominal adipose tissue
  Arms: single intra-articular injection of MM-AT

SUMMARY:
The MAST-GR study is a randomized controlled interventional trial with parallel treatment arms and 1:1 allocation

The primary objective of the study is to compare the safety and efficacy of a single intra-articular infiltration of Bone marrow aspirate concentrate (BMAC) with one of minimally manipulated adipose tissue (MM-AT) so as to determine the most effective cellular product in treating patients with knee osteoarthritis (OA).

The secondary objective is to demonstrate whether intra-articular infiltration of BMAC or MM-AT can induce disease-modifying effects in knee OA by imaging and biological assessments on peripheral blood.

The tertiary objective of the study is to identify factors that influence the clinical response to treatment (baseline characteristics of patients, biological characteristics of the treated knee, characteristics of cellular products, BMAC and MM-AT).

DETAILED DESCRIPTION:
Patients with symptomatic unilateral knee OA will be included in a randomized controlled Trial (RCT), in which one group of patients will be treated with 1 intra-articular infiltration of BMAC, and one group will be treated with 1 intra-articular infiltration of MM-AT. A total of 204 patients will be included and will undergo infiltrative treatment after collecting informed consent for study participation and master data. Patients will be clinically evaluated at 0-2-6-12 months follow-up. Possible disease-modifying effects of the two cell products will be investigated by analysis on peripheral blood at 0-2-6-12 months follow-up and by evaluation of radiographic and magnetic resonance imaging (MRI) at 0 and 12 months follow-up. In addition, characterization of the portion of BMAC and MM-AT remaining from treatment will be carried out, as well as baseline assessment of peripheral blood on all patients, and synovial fluid and synovial membrane, where possible, to analyze their influence on clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients with symptomatic unilateral knee OA with:

1. Men or women aged 40 to 75 years;
2. Signs and symptoms of OA with a clinical history of gonalgia or swelling for at least 6 months;
3. Radiographic signs of OA (Kellgren-Lawrence grade 1-4);
4. No benefit after at least 4 months of conservative treatment;
5. Ability and consent of patients to actively participate in clinical and radiological (rx and MRI) follow-up;
6. Signing of informed consent.

Exclusion Criteria:

1. Patients unable to express consent;
2. Patients aged < to 40 and > to 75 years;
3. Patients with axial deviations > 5°;
4. Patients who have suffered trauma or undergone intra-articular infiltration of other substance in the previous 6 months;
5. Patients who have undergone knee surgery in the previous 12 months;
6. Patients with concomitant knee injuries causing joint pain or swelling (-focal full-thickness osteochondral defects, acute meniscal injuries);
7. Patients with malignant neoplasms;
8. Patients with uncompensated systemic diseases (rheumatic diseases, metabolic disorders such as diabetes and thyroid diseases);
9. Patients with infectious diseases;
10. Patients with histories of alcohol or drug abuse;
11. Patients who are pregnant;
12. Patients with allergies to anesthetics used in the procedure.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster University Osteoarthritis index (WOMAC) - Pain subscale | 6 months follow-up
  It is a pathology-specific questionnaire used for the assessment of referred pain at the knee joint level in patients with OA

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 2 months, 6 months, 12 months follow-up
  It's a standardized and widely used questionnaire to assess the condition of patients with osteoarthritis of the knee and includes assessment of pain, stiffness, and physical function of the joints. It can be administered to the patient.
  It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); The score is then normalized on a 0-100 scale. Higher values indicate a worse outcome
Knee Injury and Osteoarthritis Outcome Score (KOOS) | baseline, 2 months, 6 months, 12 months follow-up
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines the following categories: symptoms, stiffness, pain, daily activities, sports and quality of life
Visual Analogue Scale (VAS) | baseline, 2 months, 6 months, 12 months follow-up
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" (0) and "the strongest pain imaginable" (10).
EuroQol Visual Analogue Scale (EQ-VAS) | baseline, 2 months, 6 months, 12 months follow-up
  EQ-VAS is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
Tegner Activity Level Scale | baseline, 2 months, 6 months, 12 months follow-up
  Tegner Activity Level Scale is a questionnaire to find out the patient's level of physical activity.All patients will indicate the type of sporting activity performed and its frequency.
Objective parameters- Range of Motion | baseline, 2 months, 6 months, 12 months follow-up
  Evaluation of the Range of Motion for comparative analysis.
Objective parameters - Circumferences | baseline, 2 months, 6 months, 12 months follow-up
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis
Patient Acceptable Symptom State (PASS) | baseline, 2 months, 6 months, 12 months follow-up
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
Minimally Clinical Important Difference (MCID) | baseline, 2 months, 6 months, 12 months follow-up
  The patient should indicate the degree of perceived improvement after the infiltrative procedure.
Expectations about the effectiveness of the treatment | baseline
  The patient should indicate at baseline what clinical benefits he or she expects from the treatment according to the question, "What benefits do you expect to get as a result of the treatment you will undergo?" the patient can choose from one of the following items:Full recovery, Definitely better, Much better, Slightly better,No change
Kellgren-Lawrence score | baseline, 12 months follow-up
  The Kellgren Lawrence scale classifies knee OA into 4 grades of subsequent greater severity, the parameters used being reduced joint space and the presence of osteophytes
3 Tesla Nuclear Magnetic Resonance Imaging (3T MRI) | baseline, 12 months follow-up
  Sequences such as T2-weighted FSE, FS-3D SPGR, and T2 Mapping will be used to assess cartilage thickness and signal, the presence of cysts and subchondral edema, joint profile, the presence of osteophytes and their size, the status of the menisci, both medial and lateral, and the status of the synovium.
Analysis of circulating micro RNAs | baseline, 2 months, 6 months, 12 months follow-up
  miRNAs, involved in OA progression, will be identified and quantified, including miR675-5p, miR-31-5p and miR-33a-5p

CONTACTS AND LOCATIONS:
Overall Officials: Luca Andriolo, MD, Principal Investigator — Istituto Ortopedico Rizzoli - II Clinica Ortopedica e Traumatologica
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
We will be able to share a subset of aggregated data, wich will not allow for the identification of participants

REFERENCES:
- [Background] Anz AW, Hubbard R, Rendos NK, Everts PA, Andrews JR, Hackel JG. Bone Marrow Aspirate Concentrate Is Equivalent to Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis at 1 Year: A Prospective, Randomized Trial. Orthop J Sports Med. 2020 Feb 18;8(2):2325967119900958. doi: 10.1177/2325967119900958. eCollection 2020 Feb. PMID 32118081
- [Background] Basile M, Rumi F, Palmeri M, Mattozzi I, Manzoli L, Mammucari M, Gigliotti S, Bernabei R, Cicchetti A. Il burden economico dell'inappropriatezza prescrittiva nella gestione dell'osteoartrite in Italia. Glob Reg Health Technol Assess. 2020 Dec 10;7:101-108. doi: 10.33393/grhta.2020.2130. eCollection 2020 Jan-Dec. Italian. PMID 36627953
- [Background] Boffa A, Merli G, Andriolo L, Lattermann C, Salzmann GM, Filardo G. Synovial Fluid Biomarkers in Knee Osteoarthritis: A Systematic Review and Quantitative Evaluation Using BIPEDs Criteria. Cartilage. 2021 Dec;13(1_suppl):82S-103S. doi: 10.1177/1947603520942941. Epub 2020 Jul 25. PMID 32713185
- [Background] Boffa A, Di Martino A, Andriolo L, De Filippis R, Poggi A, Kon E, Zaffagnini S, Filardo G. Bone marrow aspirate concentrate injections provide similar results versus viscosupplementation up to 24 months of follow-up in patients with symptomatic knee osteoarthritis. A randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2022 Dec;30(12):3958-3967. doi: 10.1007/s00167-021-06793-4. Epub 2021 Nov 12. PMID 34767030
- [Background] Cai X, Yuan S, Zeng Y, Wang C, Yu N, Ding C. New Trends in Pharmacological Treatments for Osteoarthritis. Front Pharmacol. 2021 Apr 15;12:645842. doi: 10.3389/fphar.2021.645842. eCollection 2021. PMID 33935742
- [Background] Caplan AI, Correa D. The MSC: an injury drugstore. Cell Stem Cell. 2011 Jul 8;9(1):11-5. doi: 10.1016/j.stem.2011.06.008. PMID 21726829
- [Background] Carelli S, Messaggio F, Canazza A, Hebda DM, Caremoli F, Latorre E, Grimoldi MG, Colli M, Bulfamante G, Tremolada C, Di Giulio AM, Gorio A. Characteristics and Properties of Mesenchymal Stem Cells Derived From Microfragmented Adipose Tissue. Cell Transplant. 2015;24(7):1233-52. doi: 10.3727/096368914X681603. Epub 2014 May 6. PMID 24806078
- [Background] Cavallo C, Boffa A, Andriolo L, Silva S, Grigolo B, Zaffagnini S, Filardo G. Bone marrow concentrate injections for the treatment of osteoarthritis: evidence from preclinical findings to the clinical application. Int Orthop. 2021 Feb;45(2):525-538. doi: 10.1007/s00264-020-04703-w. Epub 2020 Jul 13. PMID 32661635
- [Background] Costa V, Carina V, Conigliaro A, Raimondi L, De Luca A, Bellavia D, Salamanna F, Setti S, Alessandro R, Fini M, Giavaresi G. miR-31-5p Is a LIPUS-Mechanosensitive MicroRNA that Targets HIF-1alpha Signaling and Cytoskeletal Proteins. Int J Mol Sci. 2019 Mar 28;20(7):1569. doi: 10.3390/ijms20071569. PMID 30925808
- [Background] Costa V, Lo Dico A, Rizzo A, Rajata F, Tripodi M, Alessandro R, Conigliaro A. MiR-675-5p supports hypoxia induced epithelial to mesenchymal transition in colon cancer cells. Oncotarget. 2017 Apr 11;8(15):24292-24302. doi: 10.18632/oncotarget.14464. PMID 28061476
- [Background] Costa V, Carina V, Raimondi L, De Luca A, Bellavia D, Conigliaro A, Salamanna F, Alessandro R, Fini M, Giavaresi G. MiR-33a Controls hMSCS Osteoblast Commitment Modulating the Yap/Taz Expression Through EGFR Signaling Regulation. Cells. 2019 Nov 22;8(12):1495. doi: 10.3390/cells8121495. PMID 31771093
- [Background] Costa V, Raimondi L, Conigliaro A, Salamanna F, Carina V, De Luca A, Bellavia D, Alessandro R, Fini M, Giavaresi G. Hypoxia-inducible factor 1Alpha may regulate the commitment of mesenchymal stromal cells toward angio-osteogenesis by mirna-675-5P. Cytotherapy. 2017 Dec;19(12):1412-1425. doi: 10.1016/j.jcyt.2017.09.007. Epub 2017 Oct 27. PMID 29111380
- [Background] Costa V, De Fine M, Carina V, Conigliaro A, Raimondi L, De Luca A, Bellavia D, Salamanna F, Alessandro R, Pignatti G, Fini M, Giavaresi G. How miR-31-5p and miR-33a-5p Regulates SP1/CX43 Expression in Osteoarthritis Disease: Preliminary Insights. Int J Mol Sci. 2021 Feb 28;22(5):2471. doi: 10.3390/ijms22052471. PMID 33671114
- [Background] Durand M, Komarova SV, Bhargava A, Trebec-Reynolds DP, Li K, Fiorino C, Maria O, Nabavi N, Manolson MF, Harrison RE, Dixon SJ, Sims SM, Mizianty MJ, Kurgan L, Haroun S, Boire G, de Fatima Lucena-Fernandes M, de Brum-Fernandes AJ. Monocytes from patients with osteoarthritis display increased osteoclastogenesis and bone resorption: the In Vitro Osteoclast Differentiation in Arthritis study. Arthritis Rheum. 2013 Jan;65(1):148-58. doi: 10.1002/art.37722. PMID 23044761
- [Background] Filardo G, Perdisa F, Roffi A, Marcacci M, Kon E. Stem cells in articular cartilage regeneration. J Orthop Surg Res. 2016 Apr 12;11:42. doi: 10.1186/s13018-016-0378-x. PMID 27072345
- [Background] Filardo G, Tschon M, Perdisa F, Brogini S, Cavallo C, Desando G, Giavaresi G, Grigolo B, Martini L, Nicoli Aldini N, Roffi A, Fini M, Kon E. Micro-fragmentation is a valid alternative to cell expansion and enzymatic digestion of adipose tissue for the treatment of knee osteoarthritis: a comparative preclinical study. Knee Surg Sports Traumatol Arthrosc. 2022 Mar;30(3):773-781. doi: 10.1007/s00167-020-06373-y. Epub 2021 Jan 19. PMID 33464397
- [Background] Garza JR, Campbell RE, Tjoumakaris FP, Freedman KB, Miller LS, Santa Maria D, Tucker BS. Clinical Efficacy of Intra-articular Mesenchymal Stromal Cells for the Treatment of Knee Osteoarthritis: A Double-Blinded Prospective Randomized Controlled Clinical Trial. Am J Sports Med. 2020 Mar;48(3):588-598. doi: 10.1177/0363546519899923. PMID 32109160
- [Background] Giorgini A, Selleri F, Zambianchi F, Cataldo G, Francioni E, Catani F. Autologous micro-fragmented adipose tissue associated with arthroscopy in moderate-severe knee osteoarthritis: outcome at two year follow-up. BMC Musculoskelet Disord. 2022 Nov 8;23(1):963. doi: 10.1186/s12891-022-05921-6. PMID 36348344
- [Background] Goldring SR, Goldring MB. Changes in the osteochondral unit during osteoarthritis: structure, function and cartilage-bone crosstalk. Nat Rev Rheumatol. 2016 Nov;12(11):632-644. doi: 10.1038/nrrheum.2016.148. Epub 2016 Sep 22. PMID 27652499
- [Background] Hong Z, Chen J, Zhang S, Zhao C, Bi M, Chen X, Bi Q. Intra-articular injection of autologous adipose-derived stromal vascular fractions for knee osteoarthritis: a double-blind randomized self-controlled trial. Int Orthop. 2019 May;43(5):1123-1134. doi: 10.1007/s00264-018-4099-0. Epub 2018 Aug 14. PMID 30109404
- [Background] Iyyanki T, Hubenak J, Liu J, Chang EI, Beahm EK, Zhang Q. Harvesting technique affects adipose-derived stem cell yield. Aesthet Surg J. 2015 May;35(4):467-76. doi: 10.1093/asj/sju055. Epub 2015 Mar 18. PMID 25791999
- [Background] Jevsevar D, Donnelly P, Brown GA, Cummins DS. Viscosupplementation for Osteoarthritis of the Knee: A Systematic Review of the Evidence. J Bone Joint Surg Am. 2015 Dec 16;97(24):2047-60. doi: 10.2106/JBJS.N.00743. PMID 26677239
- [Background] Pagani S, Veronesi F, Giavaresi G, Filardo G, Papio T, Romandini I, Fini M. Autologous Protein Solution Effect on Chondrogenic Differentiation of Mesenchymal Stem Cells from Adipose Tissue and Bone Marrow in an Osteoarthritic Environment. Cartilage. 2021 Dec;13(2_suppl):225S-237S. doi: 10.1177/1947603521993217. Epub 2021 Feb 15. PMID 33583216
- [Background] Pagani S, Borsari V, Veronesi F, Ferrari A, Cepollaro S, Torricelli P, Filardo G, Fini M. Increased Chondrogenic Potential of Mesenchymal Cells From Adipose Tissue Versus Bone Marrow-Derived Cells in Osteoarthritic In Vitro Models. J Cell Physiol. 2017 Jun;232(6):1478-1488. doi: 10.1002/jcp.25651. Epub 2016 Oct 26. PMID 27739057
- [Background] Shanmugasundaram S, Vaish A, Chavada V, Murrell WD, Vaishya R. Assessment of safety and efficacy of intra-articular injection of stromal vascular fraction for the treatment of knee osteoarthritis-a systematic review. Int Orthop. 2021 Mar;45(3):615-625. doi: 10.1007/s00264-020-04926-x. Epub 2021 Jan 12. PMID 33432400
- [Background] Ulivi M, Meroni V, Vigano M, Colombini A, Lombardo MDM, Rossi N, Orlandini L, Messina C, Sconfienza LM, Peretti GM, Mangiavini L, de Girolamo L. Micro-fragmented adipose tissue (mFAT) associated with arthroscopic debridement provides functional improvement in knee osteoarthritis: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2023 Aug;31(8):3079-3090. doi: 10.1007/s00167-022-07101-4. Epub 2022 Aug 30. PMID 36040510
- [Background] Anil U, Markus DH, Hurley ET, Manjunath AK, Alaia MJ, Campbell KA, Jazrawi LM, Strauss EJ. The efficacy of intra-articular injections in the treatment of knee osteoarthritis: A network meta-analysis of randomized controlled trials. Knee. 2021 Oct;32:173-182. doi: 10.1016/j.knee.2021.08.008. Epub 2021 Sep 6. PMID 34500430
- [Background] Veronesi F, Fini M, Martini L, Berardinelli P, Russo V, Filardo G, Di Matteo B, Marcacci M, Kon E. In Vivo Model of Osteoarthritis to Compare Allogenic Amniotic Epithelial Stem Cells and Autologous Adipose Derived Cells. Biology (Basel). 2022 Apr 28;11(5):681. doi: 10.3390/biology11050681. PMID 35625409
- [Background] Veronesi F, Cadossi M, Giavaresi G, Martini L, Setti S, Buda R, Giannini S, Fini M. Pulsed electromagnetic fields combined with a collagenous scaffold and bone marrow concentrate enhance osteochondral regeneration: an in vivo study. BMC Musculoskelet Disord. 2015 Sep 2;16:233. doi: 10.1186/s12891-015-0683-2. PMID 26328626
- [Background] Veronesi F, Salamanna F, Martini L, Fini M. Naturally Occurring Osteoarthritis Features and Treatments: Systematic Review on the Aged Guinea Pig Model. Int J Mol Sci. 2022 Jun 30;23(13):7309. doi: 10.3390/ijms23137309. PMID 35806306
- [Background] Veronesi F, Desando G, Fini M, Parrilli A, Lolli R, Maglio M, Martini L, Giavaresi G, Bartolotti I, Grigolo B, Sartori M. Bone marrow concentrate and expanded mesenchymal stromal cell surnatants as cell-free approaches for the treatment of osteochondral defects in a preclinical animal model. Int Orthop. 2019 Jan;43(1):25-34. doi: 10.1007/s00264-018-4202-6. Epub 2018 Oct 15. PMID 30324310
- [Background] Veronesi F, Berni M, Marchiori G, Cassiolas G, Muttini A, Barboni B, Martini L, Fini M, Lopomo NF, Marcacci M, Kon E. Evaluation of cartilage biomechanics and knee joint microenvironment after different cell-based treatments in a sheep model of early osteoarthritis. Int Orthop. 2021 Feb;45(2):427-435. doi: 10.1007/s00264-020-04701-y. Epub 2020 Jul 14. PMID 32661637
- [Background] Veronesi F, Giavaresi G, Tschon M, Borsari V, Nicoli Aldini N, Fini M. Clinical use of bone marrow, bone marrow concentrate, and expanded bone marrow mesenchymal stem cells in cartilage disease. Stem Cells Dev. 2013 Jan 15;22(2):181-92. doi: 10.1089/scd.2012.0373. Epub 2012 Nov 16. PMID 23030230
- [Background] Veronesi F, Maglio M, Contartese D, Martini L, Muttini A, Fini M. Stromal Vascular Fraction and Amniotic Epithelial Cells: Preclinical and Clinical Relevance in Musculoskeletal Regenerative Medicine. Stem Cells Int. 2021 Feb 18;2021:6632052. doi: 10.1155/2021/6632052. eCollection 2021. PMID 33688354
- [Derived] Andriolo L, Veronesi F, Zanasi L, Costa V, Franceschini M, Miceli M, Spinnato P, Zaffagnini S, Giavaresi G, Filardo G. Adipose tissue-derived versus bone marrow-derived cell concentrates for the injective treatment of knee osteoarthritis: protocol of a prospective randomised controlled trial. BMJ Open. 2025 Apr 30;15(4):e092379. doi: 10.1136/bmjopen-2024-092379. PMID 40306987